CLINICAL TRIAL: NCT03098875
Title: Spectral Analysis of Heart Rate Variability at BIS 25 and BIS 55 Under Propofol or Sevoflurane
Brief Title: Heart Rate Variability Under Propofol and Sevoflurane
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Armand Trousseau (Other)
Responsible Party: Principal Investigator, Pr Isabelle CONSTANT, Professor, Hôpital Armand Trousseau
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HRV Propofol Sevoflurane
Record Dates: First submitted 2017-01-09; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: General Anesthesia
MeSH Terms: interventions — Sevoflurane; Propofol; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sevoflurane (Active Comparator): General anesthesia using sevoflurane as a hypnotic agent, and remifentanil as an analgesic.
  Two steady state periods of 10 minutes each, one with a steady bispectral index at 25 +/- 5, the other with a steady bispectral index at 55 +/- 5. Continuous recording of heart rate during the last minute of each steady-state. Off-line spectral analysis of heart rate variability.
  Interventions: Drug: Sevoflurane; Drug: Remifentanil
- Propofol (Active Comparator): General anesthesia using propofol as a hypnotic agent, and remifentanil as an analgesic.
  Two steady state periods of 10 minutes each, one with a steady bispectral index at 25 +/- 5, the other with a steady bispectral index at 55 +/- 5. Continuous recording of heart rate during the last minute of each steady-state. Off-line spectral analysis of heart rate variability.
  Interventions: Drug: Propofol; Drug: Remifentanil

INTERVENTIONS:
Drug: Sevoflurane — General anesthesia using sevoflurane as a hypnotic agent
  Arms: Sevoflurane
Drug: Propofol — General anesthesia using propofol as a hypnotic agent
  Arms: Propofol
Drug: Remifentanil — General anesthesia using remifentanil as an analgesic.

SUMMARY:
Patients were randomized into 2 groups according to the anesthetic, propofol or sevoflurane. Induction and maintenance were standardized, and after the end of surgery, two steady-state recordings were performed at BIS 25 and BIS 55. Bispectral Index and ECG were continuously recorded and cardiac autonomic nervous activity was investigated using spectral analysis of RR Interval variability

ELIGIBILITY:
Inclusion Criteria:

* ASA risk classification 1 or 2,
* scheduled for middle ear surgery, or cardiovascular ANS activity.

Exclusion Criteria:

* preoperative medications that interfere with the autonomic nervous system
* preoperative medications that interfere with the central nervous system

Ages: 13 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Spectral analysis of heart rate variability with a bispectral index of 25 | During surgical procedure
  Fast Fourier Transform applied to heart rate signal recording
Spectral analysis of heart rate variability with a bispectral index of 55 | During surgical procedure
  Fast Fourier Transform applied to heart rate signal recording

CONTACTS AND LOCATIONS:
Locations (1):
- Departement d'anesthesie Hopital Armand Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: No